CLINICAL TRIAL: NCT01026649
Title: The 2-stage Approach for Reducing Posterior Wall Puncture During the Internal Jugular Vein Catheterization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jae-Hyon Bahk, MD, PhD, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JHBahk_CVC two stage
Record Dates: First submitted 2009-11-19; First posted 2009-12-04 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Hematoma
Keywords: hematoma formation; success rate
MeSH Terms: conditions — Hematoma | interventions — Catheterization, Central Venous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 stage (Experimental): Approach the internal jugular vein in a 2 stage fashion during central venous catheterization
  Interventions: Procedure: Central venous catheterization
- 1 stage (Active Comparator): Approach the internal jugular vein in a traditional one stage fashion during central venous catheterization
  Interventions: Procedure: Central venous catheterization

INTERVENTIONS:
Procedure: Central venous catheterization — Approach the internal jugular vein in a traditional one stage fashion during central venous catheterization
  Arms: 1 stage
Procedure: Central venous catheterization — Approach the internal jugular vein in a 2 stage fashion during central venous catheterization
  Arms: 2 stage

SUMMARY:
To evaluate the effect of a 2-stage approach to the internal jugular vein when performing a central venous catheterization compared to the traditional one stage approach on the incidence of hematoma formation and success rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients who require a central venous catheter for their thoracic surgery

Exclusion Criteria:

* Refuse to enroll
* Infection at insertion site
* Carotid artery disease
* Anomaly of central vasculature
* Hypertrophied thyroid
* History of recent neck surgery

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2009-11; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
hematoma formation | immediately after catheterization

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea